CLINICAL TRIAL: NCT05304221
Title: Prospective Validation of the "Shamir Resistance Calculator": an Interventional Crossover Trial to Improve Empiric Prescription of Antimicrobials in Acute Care Hospitals.
Brief Title: A Prospective Cluster-Randomized, Controlled Crossover Trial to Validate an Electronic "Resistance Calculator"
Status: Recruiting | Type: Observational
Sponsor: Dror MarChaim, MD (Other Government)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor-Investigator, Dror MarChaim, MD, Head of the Unit of Infection Control & Prevention, Assaf-Harofeh Medical Center
Organization: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 0063-22-ASF
Record Dates: First submitted 2022-03-07; First posted 2022-03-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Sepsis
Keywords: MDRO; Antimicrobial Stewardship; Antimicrobial Resistance; Resistance Calculator
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Septic patients from 2 sites, who are hospitalized and require empiric antibiotic treatment, whose primary physician was assisted by the Shamir Resistance Calculator.
  Interventions: Other: Shamir Resistance Calculator
- Control group: Septic patients from 2 sites, who are hospitalized and require empiric antibiotic treatment, whose primary physician was not assisted by the Shamir Resistance Calculator.

INTERVENTIONS:
Other: Shamir Resistance Calculator — An on-line calculator which is free and accessible from all devices, which may predict the risk of MDRO infection upon admission, and the risk of nosocomial XDRO infection during the hospitalization.
  The calculator contains only parameters that could be extracted bedside, at the first presentation of a septic patient, including the ability to conduct a complete assessment also among patients with reduced consciousness and/or cognition.
  Groups: Intervention group

SUMMARY:
Primary objective:

- Our aim is to validate the "Shamir Resistance Calculator" in a prospective crossover trial, in order to shorten the time to initiation of appropriate antimicrobials among hospitalized septic patients.

Secondary objectives:

- To evaluate the impact of using the "Shamir Resistance Calculator" with regards to:

* new acquisitions of multi-drug resistant organisms (MDRO)
* the empiric usage of broad-spectrum agents (e.g., carbapenems, vancomycin)
* acute Clostridiodes difficile infections
* In-hospital mortality.

DETAILED DESCRIPTION:
2.1 List the clinical hypotheses.

* Primary hypothesis: The "Shamir Resistance Calculator" will shorten the time to initiation of appropriate antimicrobials among hospitalized septic patients.
* Secondary hypotheses: The "Shamir Resistance Calculator" will reduce the rate of new MDRO acquisitions, will reduce the empiric usage of broad-spectrum agents, will reduce the incidences of acute Clostridiodes difficile infections, and will reduce the in-hospital mortality rates among hospitalized septic patients.

2.2 Background & Rationale, Significance of Selected Topic & Preliminary Data

The world health organization (WHO) had declared that the issue of resistance to multiple antimicrobials, is one of the current and future biggest challenges and threats to human health.

* Multi-drug resistant organisms (MDRO) and extensively drug resistant organisms (XDRO) are prevalent in hospitals, in acute care settings, and also in the community.2
* The outcomes of infections caused by MDROs and XDROs are worse in comparison to susceptible organisms, mainly due to delay in initiation of appropriate antimicrobial therapy (DAAT) in those infections.3
* DAAT is the strongest independent modifiable predictor for mortality among patients with severe infections.3
* Therefore, it is of paramount importance to avoid and shorten DAAT among hospitalized septic patients.
* However, empirically prescribing unnecessary broad-spectrum agents, to patients with infections resulting from susceptible organisms, increases the burden of resistances and costs to the facility.
* Moreover, narrow-spectrum agents are frequently more potent vs. susceptible organisms (e.g., cefazolin vs. vancomycin for methicillin-susceptible Staphylococcus aureus infection4), and are frequently less toxic (e.g., colistin, vancomycin).4-6
* There are two time points, where the majority of empiric prescription errors and DAAT frequently occurs among hospitalized adults: 1) upon admission (UA) while attending patients at risk of MDRO infection, and 2) during hospitalization, while attending patients at risk of XDRO infection (MDRO are usually covered empirically in nosocomial sepsis).6
* At the first encounter with a septic patient, the primary physician needs a simple and reliable tool to be used bedside, in order to tailor an appropriate empiric antimicrobial regimen.
* Many previous attempts to develop such scores, failed to become a standard of practice, for multiple and various reasons,7-10 lacking the size and the comprehensiveness to address the whole spectrum of clinical issues and decisions.
* We developed an on-line calculator (https://assafharofe.azurewebsites.net), which is free and accessible from all devices, in order to predict the risk of MDRO infection upon admission, and the risk of nosocomial XDRO infection during the hospitalization.11
* The calculator contains only parameters that could be extracted bedside, at the first presentation of a septic patient, including the ability to conduct a complete assessment also among patients with reduced consciousness and/or cognition.
* The study that was executed in order to develop the "Shamir Resistance Calculator", which was recently published in Infection Control and Hospital Epidemiology,11 was a large study that included 4,114 patients: 2,472 patients with sepsis upon admission and 1,642 patients with nosocomial sepsis. This as far as we know, is the largest trial ever published in this field of research.
* Moreover, the calculator performances were very encouraging. The MDRO upon admission score included 10 parameters, and with a cutoff of ≥22 points, it had a ROC AUC of 0.85. The nosocomial XDRO score included 7 parameters, and with a cutoff of ≥36 points, it had a ROC AUC of 0.87.
* However, the main limitation of the on-line calculator, remains the lack of prospective data that trialed the performances of the calculator prospectively, on hard hospitalization's outcomes.
* Therefore, our goal is to trial the calculator prospectively, using the cluster randomized crossover design, which is considered today the gold standard methodology in terms of interventional studies in the field of hospital epidemiology.12

2.3 Study Design

* The study design is an interventional prospective cluster randomized crossover trial.12
* The crossover design is considered today the gold standard methodology to execute interventional trials in the field of hospital epidemiology, infection control, and antimicrobial stewardship.12 This design enables to control for multiple confounders associated with the Hawthorne effect. The intervention is implemented in same types of units. The intervention is implemented in one unit, and afterwards in the second unit, separated with washout periods prior, between, and at the end of the intervention in the second unit (i.e., to control for carryover effect of the intervention). Eventually, the independent performances of the intervention could be measured, since every unit is compared to the other unit but also the intervention period is compared to the control period in the same unit (see figure in section 2.6).
* The study will be conducted at two large Israeli acute-care hospitals: Shamir (Assaf Harofeh) Medical Center (895 beds) and Mayanei Hayeshua Medical Center (350 beds).
* Each intervention period will last 6 months and each washout period (prior to the first intervention initiation, between phases, and following the last intervention period) will last one month (see figure in section 2.6).
* The study will include all adult (>18 years) septic patients who are hospitalized and requires empiric antibiotic treatment.
* Patients with known pathogen/s for which antibiotic treatment is initiated, will not be included.
* No written informed consent will be obtained from participants, as this intervention imposes a minimal neglected potential risk to patients' safety.

  * According to Israeli regulations, these types of interventions, in the field of Infection Control / Antimicrobial Stewardship, does not necessitates obtaining written informed consent from participants. However, the protocol must be submitted, reviewed and authorized by the local IRB at both facilities, which will approve the study prior to its initiation.
  * Of note, every prescriber has the option to over-rule or ignore the calculator's results (see figure below).
  * The calculator is not aiming to replace good medical clinical judgement or practices. It is only an adjunct tool to assist physicians.
  * The calculator also serves to guide prescribers of when to involve Infectious Diseases (ID) specialist, i.e., further contributing to patient's safety.
  * The calculator has low false negative rates (14%) and excellent negative predictive value rates (98%), i.e., implying that prescribers could trustily rely on a negative result of the calculator, with high level of confidence.

2.4 Diversity & Inclusion

Diversity:

All patients above 18 years old will be included in the study. No diversity issues are relevant.

Inclusion criteria:

* Adult patients (age>18 years)
* Patients who are hospitalized at Shamir MC or at Mayanei Hayeshua MC during the study period.

  o Patients admitted to the ER and later-on discharged home, or discharged from the ER to a different facility, will be excluded as it will not enable us to follow all the designated outcomes.
* Patients for which antibiotic treatment was initiated, empirically, due to acute sepsis.

  * Patients for which antibiotics were initiated as part of a main-consolidative regimen, or as part of a pre-emptive regimen, will not be included in the study.
  * Sepsis will be defined in accordance to established criteria1.

2.7 Study Duration

The study will last 15 months (09/01/2021 - 11/30/2022).

* Study interventions are un-blinded.
* We will be able to monitor whether prescribers had used the calculator during or not during the designated intervention in their hospital, since every usage of the calculator is monitored and captured in an electronical database (i.e., this is an on-line free calculator and all results are captured and stored in secured settings).

Variables/Time Points of Interest

* Time to initiation of appropriate antimicrobials (i.e., according to the in-vitro susceptibility results of the offending isolate/s)
* New acquisitions of MDRO by patients (monitored regardless of study's purposes for Infection Control purposes).
* The amount of empiric usage of broad-spectrum agents (e.g., carbapenems, vancomycin)
* Acute C. difficile infections
* In-hospital mortality

2.8 Statistical Analysis and Sample Size Justification

Statistical Methods The performances of the calculator with regards to patients' outcomes as listed above, will be analyzed by Poisson regression models.

Power/Sample Size:

Based on our retrospective trial and preliminary data, of the patients with sepsis upon admission, 60.6% of patients with MDRO infection will suffer from DAAT for >48 hours, compared to 9.2% of patients with non-MDRO infection. This implies that at least 56 patients will need to be enrolled to each cluster (i.e., overall, 224 patients), in order to prove superiority to the intervention in 5% significance (α) and 80% power (β). Based on our preliminary retrospective trial at Shamir MC, we will expect at least ~1,000 eligible patients (i.e., patients presenting with acute sepsis for which empirical regimens are initiated) at Shamir MC during the 6-month intervention, and ~500 patients at Mayanei Hayeshua MC. Therefore, we expect the study to be way over-powered to prove the superiority of the intervention, and we plan to enroll a minimum of 120 patients for each cluster (i.e., a minimum of 480 patients overall).

2.9 Specific Drug Supply Requirements

The on-line calculator will be installed on every computer on which the electronical medical record of the facility is installed, which is used by physicians (i.e., both desktops and laptops).

2.10 Adverse Experience Reporting

AE section will be added by local PV per global templates. The investigator will act accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age>18 years)
* Patients who are hospitalized at Shamir MC or at Hadassah Medical Organization during the study period.

  o Patients admitted to the ER and later-on discharged home, or discharged from the ER to a different facility, will be excluded as it will not enable us to follow all the designated outcomes.
* Patients for which antibiotic treatment was initiated, empirically, due to acute sepsis.

  * Patients for which antibiotics were initiated as part of a main-consolidative regimen, or as part of a pre-emptive regimen, will not be included in the study.
  * Sepsis will be defined in accordance to established criteria1.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients above 18 years old will be included in the study. No diversity issues are relevant.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Time to initiation of appropriate antimicrobials. | 15 months study's period.
  The median number of days from date of enrollment to the day that the first antibiotic with in-vitro susceptibility per microbiology report was initiated.

SECONDARY OUTCOMES:
Cases of new acquisitions of MDRO by patients. | 15 months study's period.
  Amount of cases of acquisition of MDRO by naïve patients, i.e., patient was not a MDRO carrier upon admission to the index hospitalization, and became a MDRO carrier during stay.
The amount of empiric usage of broad-spectrum agents. | 15 months study's period.
  Antibiotic days of broad-spectrum agents
Acute Clostridiodes Difficile infections. | 15 months study's period.
  Incidents of new acute Clostridiodes Difficile infections.
In-hospital mortality | 15 months study's period.
  In-hospital; mortality rates

CONTACTS AND LOCATIONS:
Overall Officials: Dror MarChaim, M.D, Principal Investigator — Assaf-Harofeh Medical Center
Locations (2):
- Israel (2):
  - Shamir Medical Center (Assaf Harofeh), Be’er Ya‘aqov
  - Hadassah Medical Organization, Jerusalem

IPD SHARING:
Plan to Share IPD: No
the data is confidential and written informed consent is not obtained.

REFERENCES:
- [Background] Marchaim D, Chopra T, Bogan C, Bheemreddy S, Sengstock D, Jagarlamudi R, Malani A, Lemanek L, Moshos J, Lephart PR, Ku K, Hasan A, Lee J, Khandker N, Blunden C, Geffert SF, Moody M, Hiro R, Wang Y, Ahmad F, Mohammadi T, Faruque O, Patel D, Pogue JM, Hayakawa K, Dhar S, Kaye KS. The burden of multidrug-resistant organisms on tertiary hospitals posed by patients with recent stays in long-term acute care facilities. Am J Infect Control. 2012 Oct;40(8):760-5. doi: 10.1016/j.ajic.2011.09.011. Epub 2012 Jan 30. PMID 22285709
- [Background] Paul M, Shani V, Muchtar E, Kariv G, Robenshtok E, Leibovici L. Systematic review and meta-analysis of the efficacy of appropriate empiric antibiotic therapy for sepsis. Antimicrob Agents Chemother. 2010 Nov;54(11):4851-63. doi: 10.1128/AAC.00627-10. Epub 2010 Aug 23. PMID 20733044
- [Background] Pogue JM, Kaye KS, Cohen DA, Marchaim D. Appropriate antimicrobial therapy in the era of multidrug-resistant human pathogens. Clin Microbiol Infect. 2015 Apr;21(4):302-12. doi: 10.1016/j.cmi.2014.12.025. Epub 2015 Jan 14. PMID 25743999
- [Background] Aviv T, Lazarovitch T, Katz D, Zaidenstein R, Dadon M, Daniel C, Tal-Jasper R, Kaye KS, Marchaim D. The epidemiological impact and significance of carbapenem resistance in Pseudomonas aeruginosa bloodstream infections: a matched case-case-control analysis. Infect Control Hosp Epidemiol. 2018 Oct;39(10):1262-1265. doi: 10.1017/ice.2018.181. Epub 2018 Aug 14. PMID 30103833
- [Background] Schwaber MJ, Carmeli Y. Mortality and delay in effective therapy associated with extended-spectrum beta-lactamase production in Enterobacteriaceae bacteraemia: a systematic review and meta-analysis. J Antimicrob Chemother. 2007 Nov;60(5):913-20. doi: 10.1093/jac/dkm318. Epub 2007 Sep 11. PMID 17848376
- [Background] Marchaim D, Gottesman T, Schwartz O, Korem M, Maor Y, Rahav G, Karplus R, Lazarovitch T, Braun E, Sprecher H, Lachish T, Wiener-Well Y, Alon D, Chowers M, Ciobotaro P, Bardenstein R, Paz A, Potasman I, Giladi M, Schechner V, Schwaber MJ, Klarfeld-Lidji S, Carmeli Y. National multicenter study of predictors and outcomes of bacteremia upon hospital admission caused by Enterobacteriaceae producing extended-spectrum beta-lactamases. Antimicrob Agents Chemother. 2010 Dec;54(12):5099-104. doi: 10.1128/AAC.00565-10. Epub 2010 Sep 13. PMID 20837757
- [Background] Marchaim D, Kaye KS, Fowler VG, Anderson DJ, Chawla V, Golan Y, Karchmer AW, Carmeli Y. Case-control study to identify factors associated with mortality among patients with methicillin-resistant Staphylococcus aureus bacteraemia. Clin Microbiol Infect. 2010 Jun;16(6):747-52. doi: 10.1111/j.1469-0691.2009.02934.x. Epub 2009 Sep 11. PMID 19723135
- [Background] Tal-Jasper R, Katz DE, Amrami N, Ravid D, Avivi D, Zaidenstein R, Lazarovitch T, Dadon M, Kaye KS, Marchaim D. Clinical and Epidemiological Significance of Carbapenem Resistance in Acinetobacter baumannii Infections. Antimicrob Agents Chemother. 2016 Apr 22;60(5):3127-31. doi: 10.1128/AAC.02656-15. Print 2016 May. PMID 26883694
- [Background] Zilberman-Itskovich S, Strul N, Chedid K, Martin ET, Shorbaje A, Vitkon-Barkay I, Marcus G, Michaeli L, Broide M, Yekutiel M, Zohar Y, Razin H, Low A, Strulovici A, Israeli B, Geva G, Katz DE, Ben-Chetrit E, Dodin M, Dhar S, Parsons LM, Ramos-Mercado A, Kaye KS, Marchaim D. A "resistance calculator": Simple stewardship intervention for refining empiric practices of antimicrobials in acute-care hospitals. Infect Control Hosp Epidemiol. 2021 Sep;42(9):1082-1089. doi: 10.1017/ice.2020.1372. Epub 2021 Mar 19. PMID 33736724
- [Background] Purssell E, Drey N, Chudleigh J, Creedon S, Gould DJ. The Hawthorne effect on adherence to hand hygiene in patient care. J Hosp Infect. 2020 Oct;106(2):311-317. doi: 10.1016/j.jhin.2020.07.028. Epub 2020 Aug 5. PMID 32763330
- See also: WHO publishes list of bacteria for which new antibiotics are urgently needed. 2017 — http://www.who.int/mediacentre/news/releases/2017/bacteria-antibiotics-needed/en/.